CLINICAL TRIAL: NCT01139853
Title: Post-Operative Impact of Nasogastric Tubes on Rates of Emesis in Infants Diagnosed With Pyloric Stenosis: A Prospective, Randomized Controlled Pilot Trial
Brief Title: Post-Operative Impact of Nasogastric Tubes on Rates of Emesis in Infants Diagnosed With Pyloric Stenosis
Acronym: POINTS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POINTS
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Pyloric Stenosis
Keywords: pyloric stenosis; nasogastric tube; pyloromyotomy
MeSH Terms: conditions — Pyloric Stenosis | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasogastric Tube (Active Comparator): 10 French Nasogastric Tube inserted before surgery
  Interventions: Device: Nasogastric Tube
- No Nasogastric Tube (No Intervention)

INTERVENTIONS:
Device: Nasogastric Tube — Insertion of a 10 French Nasogastric tube prior to surgery
  Arms: Nasogastric Tube

SUMMARY:
The overall objective of this research study is to determine the effect of a pre-operatively placed nasogastric tube compared to no nasogastric tube, on post-operative emesis rates and postoperative length of stay in infants with a primary diagnosis of pyloric stenosis treated with pyloromyotomy. This study will also examine the feasibility data of the pilot data to develop estimates of treatment effect of a pre-operative nasogastric tube on post-operative rate of emesis and length of stay to be used to determine the sample size of the definitive trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infant ≤ 6 months of age
2. Primary diagnosis of Pyloric Stenosis confirmed by ultrasound
3. Amendable to circumumbilical pyloromyotomy
4. Amendable to a minimum size 10 French nasogastric tube
5. Able to undergo general anesthesia
6. Parent or legal guardian able to give free and informed consent

Exclusion Criteria:

1. Contraindicated for circumumbilical pyloromyotomy
2. Contraindicated for a size 10 French nasogastric tube
3. Prematurity before 35 weeks' gestation
4. Bronchopulmonary dysplasia
5. Viral infection in the past 7 days
6. Cardiac malformation
7. Patent ductus arteriosis
8. Previous abdominal surgery
9. Concurrent surgical procedure scheduled
10. Parent or legal guardian unable to read, speak and understand English
11. Co-enrolled in a different interventional trial

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 years

SECONDARY OUTCOMES:
post-operative length of stay | 1 year
rates of post-operative emesis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Helene Flageole, MD, FRCSC, Principal Investigator — McMaster Children's Hopsital
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Flageole HH, Pemberton J. Post-Operative Impact of Nasogastric Tubes on length of stay in infants with pyloric Stenosis (POINTS): A prospective randomized controlled pilot trial. J Pediatr Surg. 2015 Oct;50(10):1681-5. doi: 10.1016/j.jpedsurg.2015.02.023. Epub 2015 Feb 19. PMID 25783381